CLINICAL TRIAL: NCT01414881
Title: A Phase 1 Study to Assess the Effects of Mipomersen on Lipid and Lipoprotein Metabolism in Healthy Subjects
Brief Title: Study to Assess the Effects of Mipomersen on Lipid and Lipoprotein Metabolism in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: MIPO1600810
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteer
Keywords: ApoB (Apolipoprotein B); LDL (low density lipoprotein); mipomersen
MeSH Terms: interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- mipomersen (Experimental): mipomersen 200mg subcutaneously (SC) once weekly
  Interventions: Drug: mipomersen
- Placebo (Placebo Comparator): Placebo administered subcutaneously (SC) once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mipomersen — mipomersen 200mg subcutaneously (SC) once weekly
  Arms: mipomersen
Drug: Placebo — Placebo administered subcutaneously (SC) once weekly
  Arms: Placebo

SUMMARY:
The primary objective of this Phase I exploratory study is to determine the effects of mipomersen on the hepatic production of apolipoprotein-B (apo B) in very low density lipoprotein (VLDL) compared to baseline levels. The study will consist of a Screening Period, a 1-week Run-in Period to establish a stable diet, an approximate 11-week Treatment Period with Placebo or Mipomersen, and a 25-week Post-Treatment Follow-up Period. The total duration of any given subject's participation will be approximately 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating, surgically sterile, postmenopausal, abstinent, or the subject or partner is compliant with an acceptable contraceptive regimen for 4 weeks prior to Screening and willing to remain compliant with the contraceptive regimen throughout treatment and for 25 weeks after the last investigational product dose
* Body weight >50 kg, body mass index (BMI) ≤38 kg/m2, and stable weight (i.e., within 5% of mean body weight) for > 8 weeks prior to Screening
* Fasting TG levels of ≤170 mg/dL, fasting serum blood glucose of ≤115 mg/dL, and an HbA1c ≤6.5%

Exclusion Criteria:

* Presence of any clinically significant abnormal laboratory profiles, physical exams, vital signs, or ECGs
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, infectious, or psychiatric disease
* Malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for >1 year) at Screening
* History of relevant food and/or drug allergies (i.e., allergy to heparin or any significant food allergy that could preclude a stable diet)
* The subject is receiving prescription lipid-lowering therapies such as statins, bile acid sequestrants, niacin/nicotinic acid, and/or fibrates or over-the-counter (OTC) fish oils, flaxseed, red rice or nutrient supplements that might affect lipid levels
* The subject is unwilling to limit alcohol consumption for the entire duration of the study
* The subject smokes >5 cigarettes per day

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Percent change in the production rate (PR) of very low density lipoprotein (VLDL) apolipoprotein B (apo B) | through approximately 11 weeks of treatment

SECONDARY OUTCOMES:
Fractional clearance rate (FCR) of VLDL Triglyceride (TG), VLDL apo B, intermediate density lipoprotein (IDL) apo B, and low-density lipoprotein (LDL) apo B | Through approximately 11 weeks of treatment
Production rate (PR) of VLDL-TG, IDL apo B, LDL apo B | Through approximately 11 weeks of treatment
Conversion of VLDL apo B to low-density lipoprotein (LDL) apo B | Through approximately 11 weeks of treatment
Direct removal of VLDL apo B from plasma | Through approximately 11 weeks of treatment
Post-heparin hepatic lipase and lipoprotein lipase activities in serum | Through approximately 11 weeks of treatment
Fasting plasma levels of fatty acids and beta-hydroxybutyrate | Up to 40 weeks
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Columbia-Presbyterian Medical Center, MS Care Center, New York, New York, United States